CLINICAL TRIAL: NCT01888185
Title: Multimodal MRI Markers of Nigrostriatal Pathology in Parkinson's Disease
Brief Title: Identifying Biomarkers of Parkinson's Disease Using Magnetic Resonance Imaging (MRI)
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Xuemei Huang, MD, PhD, Xuemei Huang, M.D., Ph.D., Milton S. Hershey Medical Center
Other Study IDs: MSHersheyMC-40726
Record Dates: First submitted 2013-01-17; First posted 2013-06-27 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Parkinson's Disease (PD); Parkinsonism; Progressive Supranuclear Palsy (PSP); Multiple System Atrophy (MSA)
Keywords: Parkinson's; PD; nigrostriatal; substantia nigra; MRI; DTI; FA; R2*; Parkinson's Disease Biomarkers Program; PDBP; ferritin; transferrin; Fe; iron protein; PSP; MSA
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Supranuclear Palsy, Progressive; Multiple System Atrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, white blood cells, urine, cerebral spinal fluid (CSF), tissue

GROUPS / COHORTS (4):
- Parkinson's Disease (PD): Patients with a clinical diagnosis of PD (in various stages)
- Progressive supranuclear palsy (PSP): Patients with a clinical diagnosis of PSP (in various stages)
- Multiple system atrophy (MSA): Patients with a clinical diagnosis of MSA (in various stages)
- Controls: Age and gender-matched adults free from neurological disease

SUMMARY:
This study is designed to determine if magnetic resonance imaging (MRI) measures can be used to diagnose and monitor the progression of Parkinson's disease (PD) while distinguishing between PD and parkinsonisms [conditions that are PD look-a-like diseases such as progressive supranuclear palsy (PSP) or multiple system atrophy (MSA)] when combined with changes in certain proteins in body fluids that are related to iron (Fe).

DETAILED DESCRIPTION:
The lack of in vivo biomarker(s) reflecting Parkinson's disease (PD)-related cell loss and associated pathoetiological/physiological processes in nigrostriatal structures has hindered discovery research and limited the ability to evaluate disease-modifying therapies. Recent research has generated excitement for using DTI and R2* MRI measures as biomarker(s) for PD-related pathology in nigrostriatal pathways, but they fall short by the lack of understanding of their clinical implications and biological/pathological underpinnings. Working closely with the National Institute of Neurological Disorders and Stroke (NINDS) Parkinson's Disease Biomarkers Program (PDBP), the proposed work will investigate multimodal MRI techniques in combination with fluid-based iron (Fe) protein profiles to serve as in vivo markers for PD-related nigrostriatal pathology that can be used as biomarkers for diagnosing PD, following its progression, and gaining mechanistic understanding of PD pathoetiology and pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

PD Subjects:

1. Able and willing to sign the consent form at time of initial enrollment or if the subject is decisionally impaired and has a legal representative that is able and willing to sign a consent form at the time of the enrollment. If the subject becomes decisionally impaired during the course of the study, their legal representative may sign an addendum to consent for continued participation.
2. MMSE score of 15 or greater unless a legal representative is present.
3. Idiopathic PD according to published criteria.
4. History of adequate response to dopaminergic therapy.
5. History of asymmetrical symptom onset

MSA Subjects:

1. Older than 30 yrs.
2. Able and willing to sign the consent form at time of initial enrollment or if the subject is decisionally impaired and has a legal representative that is able and willing to sign a consent form at the time of the enrollment. If the subject becomes decisionally impaired during the course of the study, their legal representative may sign an addendum to consent for continued participation.
3. MMSE score of 15 or greater unless a legal representative is present.
4. MSA according to published criteria.
5. History of autonomic & urinary dysfunction and/or severe cerebellar ataxia.

PSP Subjects:

1. Older than 40 yrs.
2. Able and willing to sign the consent form at time of initial enrollment or if the subject is decisionally impaired and has a legal representative that is able and willing to sign a consent form at the time of the enrollment. If the subject becomes decisionally impaired during the course of the study, their legal representative may sign an addendum to consent for continued participation.
3. PSP according to published criteria.
4. Vertical gaze palsy and/or slow vertical gaze/postural instability during first year of diagnosis.
5. MMSE score of 15 or greater unless a legal representative is present

Controls:

1. Older than 21 yrs.
2. Able and willing to sign the consent form.
3. MMSE greater than 24.

Exclusion Criteria:

PD Subjects:

1. Unable or does not have a legal representative/unwilling to provide consent.
2. Any condition that precludes a routine MRI (e.g., claustrophobia, pacemaker, severe scoliosis, etc.).
3. History of cerebrovascular diseases or other neurological disorders.
4. Major medical problems such as renal or liver failure.
5. Unstable, non-PD-related medical conditions.
6. MMSE score less than 15 unless a legal representative is present
7. Use of anticoagulant medications.
8. Signs of dementia.

MSA Subjects:

1. Unable or does not have a legal representative /unwilling to provide consent.
2. Any condition that precludes a routine MRI (e.g., claustrophobia, pacemaker, severe scoliosis, etc.).
3. History of cerebrovascular diseases or other neurological disorders.
4. Major medical problems such as renal or liver failure.
5. Unstable, non-MSA-related medical conditions.
6. MMSE score less than 15 unless a legal representative is present
7. Use of anticoagulant medications.
8. Signs of dementia.

PSP Subjects:

1. Unable or does not have a legal representative /unwilling to provide consent.
2. Any condition that precludes a routine MRI (e.g., claustrophobia, pacemaker, severe scoliosis, etc.).
3. History of cerebrovascular diseases or other neurological disorders.
4. Major medical problems such as renal or liver failure.
5. Unstable, non-PSP-related medical conditions.
6. MMSE score less than 15 unless a legal representative is present
7. Use of anticoagulant medications.
8. Signs of dementia.

Controls:

1. Unable/unwilling to provide consent.
2. Evidence of severe memory impairment or signs of dementia (MMSE < 24).
3. Any condition that precludes a routine MRI (e.g., claustrophobia, pacemaker, severe scoliosis, etc.).
4. History of cerebrovascular diseases or other neurological disorders.
5. Major medical problems such as renal or liver failure.
6. Unstable medical conditions.
7. Use of anticoagulant medications.
8. Signs of dementia.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical patients and community volunteers
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2012-12; Primary Completion 2019-12 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Differential roles of fractional anisotropy (FA) and R2* in PD detection and progression | Change in roles of FA and R2* assessed between baseline and 18 months. Change assessed between baseline and 36 months. Change assessed between 18 and 36 months.
  Substantia Nigra (SN) FA and R2* values in PD subjects will be compared with control subjects and correlated with clinical and behavioral measures.

SECONDARY OUTCOMES:
Nigrostriatal diffusion tensor imaging (DTI) and R2* differentiate PD from parkinsonian syndromes | Assessed at baseline visit.
  DTI and R2* measures in both SN and striatal structures in PD, PSP, MSA and control subjects will be compared to assess sensitivity and specificity of individual and combined MRI measures in diagnosing PD.
Iron(Fe)-related proteins in body fluids as biomarkers of PD | Change assessed between baseline and 18 months. Change assessed between baseline and 36 months. Change assessed between 18 and 36 months.
  The protein profile in blood, urine, and cerebral spinal fluid (CSF), and their relationships to clinical and MRI measure will be interrogated with the focus being on Fe-related proteins such as hepcidin, ferritin, and transferrin.
MRI and postmortem pathological correlation | From baseline until date of death from any cause within 5 years for patient participants who succumb to their disease
  Postmortem brain analysis on patients who succumb to their disease during the study will be performed in order to inform the relationship of the biomarkers to clinical diagnosis (PD, PSP, MSA) and clinical milestones as well as to inform the pathological underpinnings of the R2* and DTI measures. In addition to standard postmortem diagnostic tests (alpha-synuclein, beta-amyloid, tau, and ubiquitin), total Fe staining, ferritin, hepcidin, tyrosine hydroxylase positive neurons, myelin and glial derived growth factors (glial cell markers) will be assessed in nigrostriatal structures in order to correlate these levels with MRI measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Milton S. Hershey Medical Center and College of Medicine, Hershey, Pennsylvania, United States

REFERENCES:
- See also: Parkinson's Disease Biomarkers Program (PDBP) description of study — https://pdbp.ninds.nih.gov/
- See also: Penn State Hershey Neurology homepage — http://www.pennstatehershey.org/web/neurology/home